CLINICAL TRIAL: NCT00595595
Title: Development of a Model to Evaluate Regenerative Endodontic Techniques
Brief Title: Development of a Model to Evaluate Regenerative Endodontic Techniques Using Extract Human Teeth
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20070149H
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Dental Pulp Regeneration; Dental Pulp Diseases
Keywords: Dental Pulp; Regenerative Medicine; Odontoblasts; Stem Cells; Growth factor differentiation of stem/progenitor cells; Odontoblast-specific cell phenotypes
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — extracted teeth 10ml of blood for DNA banking
Oversight: Data Monitoring Committee: No

SUMMARY:
Millions of teeth are saved each year by root canal therapy. Although current treatment modalities offer high levels of success for many conditions, an ideal form of therapy might consist of regenerative approaches in which diseased or necrotic pulp tissues are removed and replaced with healthy pulp tissue in order to revitalize teeth.

DETAILED DESCRIPTION:
The long term goal of this research project is to develop a method to regenerate dental pulp-like tissue as an alternative method to conventional root canal treatment. The objective of this study is to identify the methods necessary to regenerate dental pulp-like tissue in human teeth. We will collect small (~4X4mm) pieces of oral mucosa that are normally removed during surgical tooth extractions, isolate human postnatal progenitor/stem cells and, using an in vitro cell culture system, combined isolated cells with various scaffolds and test compounds to determine optimal conditions to differentiate pulp-like tissue (eg, odontoblasts, fibroblasts, endothelium, etc) grown in segments of human roots.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing indication for surgical extraction of impacted teeth
* Age 16-65

Exclusion Criteria:

* Ages less than 16 or over 65
* No pre-existing indication for surgical extraction of impacted teeth

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting for surgical removal of impacted teeth
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hargreaves, DDS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States